CLINICAL TRIAL: NCT04633382
Title: JUSTIFICATION OF THE PRINCIPLES OF ENHANCED RECOVERY AFTER BILIARY TRACT SURGERY
Brief Title: ENHANCED RECOVERY AFTER BILIARY TRACT SURGERY
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Vitebsk State Medical University (Other)
Responsible Party: Principal Investigator, Yury Arlouski, Associate professor, MD, PhD, Vitebsk State Medical University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Biliary interventional
Record Dates: First submitted 2020-11-12; First posted 2020-11-18 (Actual); Last update posted 2020-11-19 (Actual); Status verified 2020-11

CONDITIONS: Biliary Stricture; Cholangiocarcinoma; Cholangitis; Choledocholithiasis
Keywords: Fast track, Enhanced recovery after surgery, biliary surgery
MeSH Terms: conditions — Cholangiocarcinoma; Cholangitis; Choledocholithiasis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conducting research of enhanced recovery after surgery (Experimental): 1. Informing the patient about the course of the operation and the postoperative period. Psychological preparation.
  2. Refusal from complete starvation. Carbohydrate drink 2 hours before surgery.
  3. Refusal of cleansing enemas.
  4. Refusal of premedication. NSAIDs 30 minutes before surgery
  5. Prevention of thromboembolic complications
  6. Multimodal analgesia: epidural catheter, paracetamol.
  7. Minimally invasive access.
  8. Prevention of hypothermia
  9. Targeted infusion therapy.
  10. Failure or limited time use of drainages: gastric, intra-abdominal, bile duct drainage.
  11. Early activation of the patient.
  12. Early enteral nutrition.
  13. Prevention of nausea and vomiting.
  Interventions: Combination Product: Enhanced recovery after biliary tract surgery
- Conducting research of traditional recovery after surgery (Placebo Comparator): 1. Informing the patient about the course of the operation and the postoperative period. Psychological preparation.
  2. Fasting for 2 days
  3. Use of cleansing enemas. Bowel preparation
  4. Premedication
  5. Prevention of thromboembolic complications
  6. Without multimodal analgesia
  7. Traditional access.
  8. Prevention of hypothermia
  9. Targeted infusion therapy.
  10. Use of drains: gastric, intra-abdominal, bile duct drainage.
  11. Activation of patients within 2 days.
  12. Enteral nutrition after 2 days after surgery.
  13. Without the use of metoclopramide
  Interventions: Combination Product: Enhanced recovery after biliary tract surgery

INTERVENTIONS:
Combination Product: Enhanced recovery after biliary tract surgery — Patients with malignant and benign diseases of the bile ducts, who have formed various types of anastomosis in two options for managing the postoperative period: traditional and based on the principles of enhanced recovery after surgery

SUMMARY:
The aim of the study is to improve the immediate results after reconstructive and restorative operations on the biliary tract by substantiating the management of the perioperative period on the principles of "enhanced recovery after surgery".

DETAILED DESCRIPTION:
A prospective randomized study on the effect of fast-track surgery on the immediate postoperative results after various reconstructive and restorative operations on the bile ducts. In the Department of Surgical Hepatology and Transplantation, a prospective randomized study will include patients (about 50) with planned reconstructive and restorative operations on the bile ducts for malignant and benign diseases of the bile ducts.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with malignant diseases of the biliary tract (cholangiocarcinoma):

   1.1. tumor resectability 1.2. absence:
   * distant metastases
   * carcinomatosis
   * perforation of the tumor and peritonitis
   * sprouting into adjacent organs and tissues (locally advanced cancer)
   * total adhesion process in the abdominal cavity (after previous operations). 1.3. Planned reconstructive surgery on the biliary tract.
2. Patients with benign biliary tract pathology. 2.1. Planned reconstructive or restorative surgery on the biliary tract for the following diseases:

   * choledocholithiasis
   * Mirizzi syndrome
   * cysts of the common bile duct
   * strictures of the common bile duct
   * injuries to the bile ducts
   * adenoma and stricture of the OBD

Exclusion Criteria:

1. Scale ASA> III (severe concomitant cardiovascular pathology).
2. Palliative reconstructive surgery.
3. Previously performed operations on the bile ducts (up to 1 month).
4. Cachexia.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-01-01 (Estimated); Primary Completion 2021-01-31 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
Reduction of bed-days | 1 week
  Improvement of basic health indicators, absence of complications, reduction of bed days

IPD SHARING:
Plan to Share IPD: No